CLINICAL TRIAL: NCT06624202
Title: COmmunities Aligned to Reduce Concussion and Head Impact Exposure (COACH)
Brief Title: COmmunities Aligned to Reduce Concussion and Head Impact Exposure
Acronym: COACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00119368; R01HD116966 (NIH)
Record Dates: First submitted 2024-10-01; First posted 2024-10-02 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Concussions
Keywords: football injuries; subconcussive head impacts; head impact exposure
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Biomechanical data collection will occur during youth football practices and games.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- practice intervention (Experimental): head impact outcomes will be monitored from athletes enrolled on teams participating in the COmmunities Aligned to reduce Concussion and Head impact exposure (COACH) intervention
  Interventions: Behavioral: COmmunities Aligned to reduce Concussion and Head impact exposure (COACH) Intervention

INTERVENTIONS:
Behavioral: COmmunities Aligned to reduce Concussion and Head impact exposure (COACH) Intervention — COmmunities Aligned to reduce Concussion and Head impact exposure (COACH) includes use of practice plans and a resource booklet aligned with the National Federation for High School guidelines for contact in practice. Coaches will also attend a pre-season coaches' clinic and be paired with a peer mentor during the season.

SUMMARY:
Head impacts in collision sports such as football are a public health concern, as repetitive head impacts, even if a concussion is not suspected, have negative effects on brain health. This study has partnered with a community stakeholder group to create a safety program for youth football named "COmmunities Aligned to reduce Concussion and Head impact exposure (COACH)", which seeks to improve knowledge and skills of youth coaches in effective and safe practice planning and to change attitudes and beliefs to prevent head impacts and promote safety. To continue advancing COACH as an approach to prevent head injuries in youth football, this R01 Research Project Grant will determine the ability of youth football organizations to adopt COACH and test if COACH is effective in reducing head impacts, concussion, and negative effects of brain health while monitoring how the program is implemented.

DETAILED DESCRIPTION:
Football has a high risk of concussion and incidence of subconcussive head impacts which have long-lasting negative effects on brain health. With roughly 3.5 million athletes participating in youth football each year, there is a critical need to reduce head impact exposure and concussion risk. Over an entire season, most of an athlete's head impact exposure is attributed to practice. Coach-directed activities (e.g., practice drills) influence the frequency and severity of head impact exposure. Practices are amenable to intervention; however, youth football leagues are often community-run organizations with limited resources, making implementation and enforcement of injury prevention strategies a challenge. Thus, engaging community members is essential for successful development, implementation, and sustenance of interventions. This study partnered with a community stakeholder group to co-design and implement an evidence-based intervention program: COmmunities Aligned to reduce Concussion and Head impact exposure (COACH). COACH seeks to improve knowledge and skills of youth football coaches in effective practice planning that incorporates safe drills and to change attitudes and beliefs toward contact in practice. COACH has been pilot tested in two teams and shown to be acceptable and feasible. A critical next step of this research is the pragmatic evaluation of the effectiveness of COACH on a larger scale, while identifying factors that influence implementation. This study addresses this critical next step by determining the capacity of youth football organizations to adopt COACH and by testing COACH's effectiveness while monitoring the implementation process.

ELIGIBILITY:
Inclusion Criteria:

* Participants without braces

Exclusion Criteria:

* Athletes will be excluded from participation if they currently have braces or plan to have braces during the football season, or have dental appliances that may impede the fit of the mouthpiece device (e.g., Herbst Appliance).

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 880 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of practice impacts | 3 months
  Total number of head impacts measured during the season in practices - 0-500 impacts
linear acceleration of practice impacts | 3 months
  Median peak resultant linear acceleration measured during the season in practices - 8-45 g of linear acceleration
rotational acceleration of practice impacts | 3 months
  Median peak resultant rotational acceleration measured during the season in practices - Median peak resultant linear acceleration measured during the season in practices - 8-45 g of linear acceleration - 100-1500 rad/s^2
Change in verbal memory composite (ImPACT) scores | 3 months
  Pre- to post-season change in attentional processes, learning, and memory within the verbal domain - range: 60-100; The composite score represents the average performance across three subtasks. A higher score indicates better performance.
Change in visual memory composite (ImPACT) scores | 3 months
  Pre- to post-season change in visual attention and scanning, learning, and memory - range :40-100 The composite score represents the average performance across two subtasks. A higher score indicates better performance.
Change in visual motor speed composite (ImPACT) scores | 3 months
  Pre- to post-season change in visual processing, learning and memory, and visual-motor response speed - range: 20-50 The composite score represents the average performance across two subtasks. A higher score indicates better performance.
Change in reaction time composite (ImPACT) scores | 3 months
  Pre- to post-season change in response speed - range: 0-1; The composite score represents the average performance across three subtasks. A lower score indicates better performance.
Change in Flanker Task (NIH Toolbox) Scores | 3 months
  Pre- to post-season change in inhibitory control and attention; range: 0-10 - Scoring is based on a combination of accuracy and reaction time. A higher score indicates better performance.
Change in pattern comparison (NIH Toolbox) Scores | 3 months
  Pre- to post-season change in processing speed; range: 0-130 - Raw score is the number of items correctly in 85 seconds; score is then converted to a normative standard score. A higher score indicates better performance.
Change in list sorting (NIH Toolbox) Scores | 3 months
  Pre- to post-season change in working memory; range: 0-26 - Scored by summing the total number of items correctly recalled and sequenced, then converted to a nationally normed score. A higher score indicates better performance.
Change in Postural Control Scores | 3 months
  participants will complete two 30-second trials (one with eyes opened, one with eyes closed).
  Five measurements will be calculated at each time point (pre- and post-season): anterior-posterior sway, medial-lateral sway, path length, maximum path velocity, and center of pressure area.
Change in Conners' Continuous Performance Test (CPT) Scores | 3 months
  Participants will complete a 14-minute computer-based assessment that evaluates selective, sustained and divided attention, as well as impulsivity and vigilance - If the T-score is below 60, it is usually unlikely that the individual has ADHD. A score above 60 might suggest Attention-deficit/hyperactivity disorder (ADHD), and if it's over 70, it could indicate more serious symptoms. Scores ranging from 0-177 with higher scores denoting more symptoms

SECONDARY OUTCOMES:
Intervention fidelity percentage of implementation | 3 months
  Implementation score representing the percentage of practices the intervention was implemented as prescribed - 0-100% - higher percent denoting more implementation
Adaptation of the intervention (AIM) score | pre-season
  5-point Likert scale of the acceptability of the intervention - 0-5 - higher scores denoting more adaptation
Feasibility of the Intervention (FIM) score | pre-season
  5-point Likert scale of the feasibility of the intervention - 0-5 - higher scores denoting higher feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Urban, PhD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data that underlie the primary outcomes reported in papers after deidentification
Supporting Information: Study Protocol, SAP
Time Frame: 6 months After Publication
Access Criteria: Researches who provide a methodologically sound proposal; to achieve the aims of the approved proposal